CLINICAL TRIAL: NCT04333407
Title: Preventing Cardiac Complication of COVID-19 Disease With Early Acute Coronary Syndrome Therapy: A Randomised Controlled Trial.
Acronym: C-19-ACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting eligible participants
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20HH5868
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: Coronavirus, SARS-CoV-2, COVID-19, Cardiovascular
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Aspirin; Clopidogrel; Rivaroxaban; Atorvastatin; Omeprazole

STUDY DESIGN:
Intervention Model Description: Prospective Multicentre Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental)
  Interventions: Drug: Aspirin 75mg; Drug: Clopidogrel 75mg; Drug: Rivaroxaban 2.5 MG; Drug: Atorvastatin 40mg; Drug: Omeprazole 20mg
- Control Arm (No Intervention)

INTERVENTIONS:
Drug: Aspirin 75mg — • If patient not on aspirin, add aspirin 75mg once daily unless contraindicated.
  Arms: Active Arm
Drug: Clopidogrel 75mg — • If patient not on clopidogrel or equivalent, add clopidogrel 75mg once daily unless contraindicated
  Arms: Active Arm
Drug: Rivaroxaban 2.5 MG — * If patient not on an anticoagulation, add rivaroxaban 2.5mg bd unless contraindicated
  * If patient on DOAC then change to rivaroxaban 2.5mg unless contraindicated
  Arms: Active Arm
Drug: Atorvastatin 40mg — • If patient not on a statin, add atorvastatin 40mg once daily unless contraindicated
  Arms: Active Arm
Drug: Omeprazole 20mg — • If patient not on a proton pump inhibitor, add omeprazole 20mg once daily.
  Arms: Active Arm

SUMMARY:
The outbreak of a novel coronavirus (SARS-CoV-2) and associated COVID-19 disease in late December 2019 has led to a global pandemic. At the time of writing, there have been 150 000 confirmed cases and 3500 deaths. Apart from the morbidity and mortality directly related to COVID-19 cases, society has had to also cope with complex political and economic repercussions of this disease.

At present, and despite pressing need for therapeutic intervention, management of patients with COVID-19 is entirely supportive. Despite the majority of patients experiencing a mild respiratory illness a subgroup, and in particular those with pre-existing cardiovascular disease, will experience severe illness that requires invasive cardiorespiratory support in the intensive care unit.

Furthermore, the severity of COVID-19 disease (as well as the likelihood of progressing to severe disease) appears to be in part driven by direct injury to the cardiovascular system. Analysis of data from two recent studies confirms a significantly higher likelihood of acute cardiac injury in patients who have to be admitted to intensive care for the management of COVID-19 disease.

The exact type of acute of cardiac injury that COVID-19 patients suffer remains unclear. There is however mounting evidence that heart attack like events are responsible. Tests ordinarily performed to definitely assess for heart attacks will not be possible in very sick COVID-19 patients. Randomising patients to cardioprotective medicines will help us understand the role of the cardiovascular system in COVID-19 disease. It will also help us determine if there is more we can do to treat these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19 infection
2. Age =/>40 or diabetes or known coronary disease or hypertension
3. Requires hospital admission for further clinical management.

Exclusion Criteria:

1. Clear evidence of an acute coronary syndrome or myo-pericarditis that requires specific treatment that precludes randomization.
2. Evidence of active bleeding
3. Pregnancy.
4. Age <18 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  All-cause mortality

SECONDARY OUTCOMES:
An ordinal outcome measure of 4 levels (1 - Death, 2 - Intensive Care Unit environment, 3 - In Hospital, 4 - At Home). | 30 days
  - In Hospital, 4 - At Home), using a Bayesian longitudinal ordinal model over 30 days
Peak troponin | 7- and 30- days
  Peak troponin within 7- and 30-days post randomization, if available.
Time to discharge | Up to 30 days
  Time to hospital discharge (length of stay)
Need for non-invasive ventilatory support | 30 days
  Need for non-invasive ventilatory support, if data available.
Need for invasive ventilatory support | 30 days.
  Need for invasive ventilatory support, if data available.
Need for mechanical circulatory support | 30 days
  Need for mechanical circulatory support, if data available.
Need for renal replacement therapy | 30 days
  Need for renal replacement therapy, if data available.
Bleeding Academic Research Consortium (BARC) bleed event | 30 days
  Bleeding Academic Research Consortium (BARC) bleed event, adjudicated
Cessation of randomized active arm therapy | 30 days
  Cessation of randomized active arm therapy

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, FRCP, PhD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers or organisations. Anonymised data might be shared with other research organisations